CLINICAL TRIAL: NCT00467597
Title: Quantification of Levodopa Induced Dyskinesia in Parkinson Disease: Developing Objective Measures of Levodopa Induced Dyskinesia (Study One)
Brief Title: Developing Objective Measures of Levodopa Induced Dyskinesia: (Study 1)
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: RCD-003-05F
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Dyskinesias; Movement Disorders; Parkinson Disease
Keywords: Dyskinesia; Levodopa; Movement Disorders; Parkinson Disease
MeSH Terms: conditions — Dyskinesias; Movement Disorders; Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Levodopa (delivered intravenously)

INTERVENTIONS:
Drug: Levodopa (delivered intravenously) — IV Levodopa is given from 09:00 to 11:00 am during the testing phase of the study. The IV Levodopa allows the researchers to watch one full "on" and "off" levodopa cycle while in the inpatient unit.

SUMMARY:
The ultimate goal of this proposal is to reduce dyskinesia in Parkinson's Disease (PD) patients. Dyskinesias are abnormal movements, often caused by the standard treatment for PD symptoms, levodopa. In this study, we will test if biochemical devices are equal to the clinical rating system in measuring dyskinesias.

DETAILED DESCRIPTION:
Levodopa induced dyskinesia (LID) is a major problem associated with chronic use of levodopa (LD) for symptomatic treatment of Parkinson's disease (PD). LD remains our most potent therapy and nearly all PD patients will use it. A substantial portion of them will experience LID, with the impact ranging from non-interfering to severely disabling. The objective of this study is to develop reliable and sensitive objective measures of LID that will quantify muscular control and postural stability in subjects with dyskinesia.

While the "gold standard" of measuring LID is the subjective RS, we will determine if objective biochemical devices will equal the reliability and validity of CRS. We hypothesize that force plate technology quantifies postural sway movements best, and pinch-grip will best quantify muscle overflow force during voluntary movements.

We will compare two biomechanical devices and a traditional clinical rating scale (CRS). Once biomechanical instrument measures LID in the setting of voluntary muscle activity, the other acquires LID data related to postural sway.. A cross-section of LD-treated patients with and without clinically apparent dyskinesia will be used to assess the measures.

32 subjects will be invited to participate, 24 with PD and 8 age-matched controls (likely unaffected spouses) without neurologic disease. Of the PD patients 7 will have no clinically apparent dyskinesia, 7 will have mild dyskinesia and 7 with moderate to severe dyskinesia will be recruited (3 additional subjects are included to account for missing data or drop-outs).

They will comfortably stand with their feet placed in a preset marked stance on the force plate either with or without a mental task and pick up a pinch-grip device multiple times. Testing will be done in the effective motor "on" and "off" states to establish validity and reliability of instrument data, as these states often reflect the usual clinical experience of patients. The second method for rating dyskinesia will be the Clinical Rating Scale. Subjects will be rated while standing on the force plate during both mental task and non-mental task conditions.

All subjects will undergo this testing. Healthy subjects will undergo this testing three times during one visit. Subjects with PD will be admitted overnight, and have seven testing periods which will vary in the number of times the procedures will be done. Inpatient subjects will also receive 1mg/kg/hr or 1.5mg/kg/hr of intravenous levodopa depending on their everyday usage of levodopa or levodopa equivalent medications for 2 hours (9AM - 11AM) with carbidopa 25 mg po at 8AM, 10AM and noon to prevent nausea.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable idiopathic Parkinson's Disease or no neurologic disease (no disease for controls only)
* At least 21 years of age
* Mini Mental Status Exam Score>=25

Exclusion Criteria:

* Evidence of psychosis (hallucinations or delusions) by history
* Any unstable medical condition
* Currently using dopamine blocking medication
* Currently taking anticoagulants or MAO inhibitors

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients on Levodopa with or without dyskinesia (abnormal involuntary movements caused by levodopa usage).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2006-04; Primary Completion 2008-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Anne Chung, MD, Principal Investigator — VA Medical Center, Portland
Locations (1):
- VA Medical Center, Portland, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Parkinson's Disease: Parkinson's disease with and without Levodopa-Induced Dyskinesia (no intervention).
- Controls: Non-Parkinson's Disease Controls (no intervention).
Period: Overall Study
Arm/Group | Parkinson's Disease | Controls
Started | 26 | 6
Completed | 24 | 6
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- PD - No LID: Parkinson's disease without levodopa-induced dyskinesia
- PD - Mild LID: Parkinson's disease with mild to moderate levodopa-induced dyskinesia (mAIMS <= 7)
- PD - Mod LID: Parkinson's disease with moderate to severe levodopa-induced dyskinesia (mAIMS > 8)
- Controls - No PD: Controls with no Parkinson's disease
- Total: Total of all reporting groups
Arm/Group | PD - No LID | PD - Mild LID | PD - Mod LID | Controls - No PD | Total
Number analyzed (Participants) | 6 | 11 | 4 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (6.1) | 62.8 (10.6) | 61.4 (6.8) | 68.3 (8.2) | 64.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 5 | 10 | 3 | 5 | 23
Region of Enrollment [Number; unit: participants]
  United States | 6 | 11 | 4 | 6 | 27
Duration of Disease (years) [Mean (Standard Deviation); unit: years] | 4.7 (3.1) | 10.2 (5.0) | 10.5 (4.8) | 0 (0) | 9.5 (5.9)
UPDRS (part III) [Mean (Standard Deviation); unit: units on a scale] — Unified Parkinson's Disease Rating Scale - Part III (Motor Section). This scale rates from 0 (normal) to 4 (Can barely perform the task) several motor areas including speech, facial expression, tremor, rigidity, hand movements, agility, posture, and gait. Higher values on this scale represent a more severe stage of the disease. the total score ranges from 0 to 108, with higher scores representing a more sever stage of the disease.
  units on a scale | 21.3 (7.9) | 23.5 (12.7) | 12.0 (8.0) | 0 (0) | 15.3 (13.1)
mAIMS at Screening [Mean (Standard Deviation); unit: units on a scale] — Modified Abnormal Involuntary Movement Rating Scale (mAIMS). This is a commonly utilized scale that is completed by an observer who judges the severity of levodopa induced dyskinesia (LID) in 7 body parts (face, neck, trunk, both legs, and both arms) during the finger tapping task, and during the Get-Up and go task (both described below). All body parts are rated separately on this 0 (none) to 4 (severe - markedly impairs activities) scale. Thus, the total score can range from 0 - 28 with 28 indicating the most severe LID.
  units on a scale | 0 (0) | 1.6 (2.4) | 11.8 (3.5) | 0 (0) | 3.1 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Gaitmat Stance Measurements (AUC)
Description: Gaitmat stance measurements were measured every half hour throughout an 8 hour period. Area under the curve was computed using the trapezoidal method for root mean squared velocity in the anterior-posterior direction. Each subject's unique baseline was used by computing the mean of the test-retest period measured at 08:00 am.
Time Frame: Every 1/2 hour during an 8 hour period.
Measure: Mean (Standard Deviation); unit: Root Mean Square of Velocity*Minutes
Arm/Group | PD - No LID | PD - Mild LID | PD - Mod LID | Controls - No PD
Number analyzed (Participants) | 6 | 11 | 4 | 6
Root Mean Square of Velocity*Minutes | 4.48 (2.1) | 10.8 (12.1) | 20.9 (26.0) | 2.8 (0.95)

ADVERSE EVENTS:
Arm/Group | PD - No LID | PD - Mild LID | PD - Mod LID | Controls - No PD
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/11 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/11 | 0/4 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes